CLINICAL TRIAL: NCT03590106
Title: Cardiac Surgery Peer Recovery Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, David Goede, Clinical Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SON2018-001; NCT03642379 (obsolete NCT alias)
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: IV Drug Usage; Infective Endocarditis; Substance Use Disorders
MeSH Terms: conditions — Endocarditis; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: All patients meeting the eligibility criteria will be approached about participation in the Peer Recovery Support Program. Those who agree will receive the intervention as designed. Those who receive will continue to receive standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Recovery Support Program (Experimental): Patients enrolled in the Peer Recovery Support Program will:
  1. Actively engage in the program as defined by meeting with a Peer Support Volunteer at least two times prior to discharge, and or use of resilience journal, and or review of NA book.
  2. Demonstrate negative drug screens done randomly during their hospitalization.
  3. Actively contact at least one outpatient recovery program that they might enroll in prior to discharge (information about recovery programs to be provided by unit SW).
  4. Demonstrate appropriate changes in their SOCRATES 8D survey scores from admission to program to post discharge.
  5. Participate in follow up phone call with completion of SOCRATES 8D survey at 30 and 60 days post discharge.
  Interventions: Behavioral: Peer Recovery Support Program

INTERVENTIONS:
Behavioral: Peer Recovery Support Program — See above

SUMMARY:
The purpose of the study is to develop and implement an addiction recovery support program for cardiac surgery patients admitted with a diagnosis of infective endocarditis secondary to IV drug addiction.

This is a single center/single unit (7-3600) exploratory study to examine the efficacy of three interventions on a subject's SOCRATES 8D score at time of discharge, at three months, and at six months. A convenience sample of all patients admitted to 7-3600 who meet the inclusion criteria for this study will be approached and provided information related to this study. Once entered into the study, the subjects will continue in the study through their hospitalizations and up to 60 days post hospitalization.

This is a quality improvement study designed specifically for the cardiac surgery population. The unit is the primary unit that subjects who are admitted with IE are located. The study's objectives include:

By date of discharge, subjects enrolled in the Peer Recovery Support Program will:

1. Actively engage in the program as defined by meeting with a Peer Support Volunteer at least two times prior to discharge, and or use of resilience journal, and or review of NA book.
2. Demonstrate negative drug screens done randomly during their hospitalization.
3. Actively contact at least one outpatient recovery program that they might enroll in prior to discharge (information about recovery programs to be provided by unit SW).
4. Demonstrate appropriate changes in their SOCRATES 8D survey scores from admission to program to post discharge.
5. Participate in follow up phone call with completion of SOCRATES 8D survey at 30 and 60 days post discharge.

DETAILED DESCRIPTION:
In 2015, Cardiac Surgery service at the University of Rochester Medical Center surgically treated 33 patients with IE. Of these 33, 12 patients had a history of IV drug use prior to their admission. Five patients had recent IV drug use which is defined as use less than 30 days prior to admission. In 2016, Cardiac Surgery service surgically treated 41 patients with endocarditis. Of these 41, 20 patients had a history of recent IV drug use prior to their admission. Nine patients had recent IVDU. In 2017, IE admissions did decrease, 16 patients with IE were surgically treated. Of these, 6 patients had recent IVDU prior to admission (Figure 3) (P. Krause, personal communication, 12/20/2017). These numbers only represent the patients that had undergone surgical repair/replacement of their cardiac valves and thus do not include the patients that were admitted to the cardiac surgery service, medically managed, and then transferred or discharged to home.

The investigators do not have a total number of target subjects due to the variability of admissions with IE. The goal is to have at least 10 subjects enrolled and complete all follow ups.

1. Inclusion Criteria:

   All patients considered for this program must meet the following criteria:
   1. Must be at least 18 years of age and able to provide consent
   2. Must speak/read/understand English
   3. Currently hospitalized and physically located on 7-3600 unit
   4. Followed by or on the Cardiac Surgery service
   5. Have a diagnosis of Endocarditis associated with recent or remote intravenous drug use (IVDU)
   6. Alert and oriented to person, place, time, and events leading up to hospitalization
   7. Able to carry on a coherent conversation
   8. Clinical Opiate Withdrawal (COW) score of less than or equal to 5 with no adjunctive (opioids) medication use within past 24 hours a. If COW score is greater than five or adjunctive medications have been used within the previous 24 hours, the patient will be re-evaluate every 24 hours until score is less than or equal to five and no adjunctive medications used within the previous 24 hours
2. Exclusion Criteria:

   1. Under the age of 18 years old
   2. Unable to speak/read/understand English
   3. Hospitalized but not on 7-3600
   4. Does not have a diagnosis of endocarditis associated with IVDU
   5. Not followed by or on the Cardiac Surgery service
   6. Not Alert or oriented or unable to carry on a coherent conversation
   7. COW score that is greater than five or adjunctive medications have been used within the previous 24 hours (see inclusion criteria)

ELIGIBILITY:
Inclusion Criteria:

All patients considered for this program must meet the following criteria:

1. Must be at least 18 years of age and able to provide consent
2. Must speak/read/understand English
3. Currently hospitalized and physically located on 7-3600 unit
4. Followed by or on the Cardiac Surgery service
5. Have a diagnosis of Endocarditis associated with recent or remote intravenous drug use (IVDU)
6. Alert and oriented to person, place, time, and events leading up to hospitalization
7. Able to carry on a coherent conversation
8. Clinical Opiate Withdrawal (COW) score of less than or equal to 5 with no adjunctive (opioids) medication use within past 24 hours a. If COW score is greater than five or adjunctive medications have been used within the previous 24 hours, the patient will be re-evaluate every 24 hours until score is less than or equal to five and no adjunctive medications used within the previous 24 hours

Exclusion Criteria:

1. Under the age of 18 years old
2. Unable to speak/read/understand English
3. Hospitalized but not on 7-3600
4. Does not have a diagnosis of endocarditis associated with IVDU
5. Not followed by or on the Cardiac Surgery service
6. Not Alert or oriented or unable to carry on a coherent conversation
7. COW score that is greater than five or adjunctive medications have been used within the previous 24 hours (see inclusion criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
SOCRATES 8D | 60 days post-discharge
  Personal Drug Use Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Goede, DNP ACNP-BC, Principal Investigator — University of Rochester School of Nursing
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No